CLINICAL TRIAL: NCT00880256
Title: Mindfulness-Based Stress Reduction for Bowel Symptoms: Collection of Pilot Survey Data
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Responsible Party: Principal Investigator, David Kearney, Staff Physician,, Seattle Institute for Biomedical and Clinical Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0013
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel; mindfulness; stress; meditation
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MBSR (Experimental): Patients who undergo mindfulness-based stress reduction will fill out measures of IBS severity before and after the mindfulness course.
  Interventions: Behavioral: mindfulness-based stress reduction

INTERVENTIONS:
Behavioral: mindfulness-based stress reduction — An 8-week course in mindfulness training

SUMMARY:
Irritable bowel syndrome (IBS) is a very common, chronic disorder that significantly affects quality of life, and results in enormous expenditures each year in the United States. Therapy for IBS is generally unsatisfactory, and takes an additive approach whereby medications are prescribed according to each type of symptom the patient experiences. Accumulating evidence indicates that persons with IBS have a heightened perception of stress, and chronic stress has been shown to have a significant impact on IBS symptomatology. Mindfulness involves the ability to bring attention to the present moment without judgment; this ability is correlated with measures of mental health and decreased stress perception. The clinical literature suggests that mindfulness-based interventions may lead to improvement in many disorders including chronic pain, stress, anxiety, eating disorders and depressive relapse. The purpose of this study is to collect survey pilot data to determine whether an 8-week program of mindfulness-based stress reduction (MBSR) improves symptoms and quality of life for persons with IBS. Patients in the 8-week MBSR program are referred as part of their clinical care, and we seek approval only to collect survey data before and after the MBSR course. This study will evaluate whether there is sufficient evidence of efficacy to warrant a full clinical trial of MBSR.

DETAILED DESCRIPTION:
Aim 1: Apply measures of IBS symptom severity, depression and quality of life before and after the MBSR course, to assess whether there is evidence of benefit, and allow calculation of standardized effect sizes. Aim 2: Apply a validated measure of mindfulness before and after treatment. Aim 3: Explore the relationship between IBS symptoms, mindfulness score, and frequency of mindfulness practice.

ELIGIBILITY:
Inclusion Criteria:

* All patient who enroll in a MBSR course

Exclusion Criteria:

* Psychosis, borderline personality, active substance abuse

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2008-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kearney, MD, Principal Investigator — VA Puget Sound Heatlh Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During a 17-month period, we enrolled 93 patients who were referred or self-referred themselves to the Mindfulness-Based Stress Reduction (MBSR) program at VA Puget Sound.
Period: Overall Study
Arm/Group | MBSR
Started | 93
Completed | 65
Not Completed | 28
Not completed — Lost to Follow-up | 28

BASELINE CHARACTERISTICS:
Arm/Group | MBSR
Number analyzed (Participants) | 93
Age Continuous [Mean (Standard Deviation); unit: years] | 51 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 69

OUTCOME MEASURES:

1. Primary Outcome: IBS (Irritable Bowel Syndrome) Symptom Severity Score (Total Score)
Description: The Irritable Bowel Severity Scoring System (IBSSS) provides a measure of the severity of IBS. The measure consists of five questions, which assess severity of abdominal pain, number of days with abdominal pain in past 10 days, severity of abdominal distension, satisfaction with bowel habits, and impact of IBS on life in general. The score on each of the 5 questions ranges from 0 to 100, and the scores are summed with a range of total possible scores from 0 to 500. Higher scores reflect more severe IBS. Total score was used in the analyses.
Time Frame: 6 months
Population: We compared scores at baseline, 2-month, and 6-month time points, using t-tests. A two-sided P value of less than 0.05 was considered statistically significant. The standardized mean difference (Cohen's d effect size) from baseline to 2-months, and baseline to 6-months was calculated for each variable.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mindfulness-Based Stress Reduction (MBSR): Patients who undergo mindfulness-based stress reduction will fill out measures of IBS severity before and after the mindfulness course.
Arm/Group | Mindfulness-Based Stress Reduction (MBSR)
Number analyzed (Participants) | 65
units on a scale
  IBS (IBS) symptoms | 256.9 (90.6)
  Irritable Bowel Syndrome Quality of LIfe (QOL) | 84.4 (20.6)

2. Secondary Outcome: Irritable Bowel Syndrome (IBS) Quality of Life
Description: The IBS-QOL is a disease specific Quality-of-Life Measure for IBS. IBS-QOL has been shown have a high level of content validity and to be responsive to change, and has been used in several outcome studies and clinical drug trials throughout the world. It consists of 34 questions that assess the influence of bowel habits on daily life. The response to each question is rated on a 5-point scale. A lower score indicates worse bowel-related quality of life. The summed total score is transformed to a 0-100 scale ranging from 0 (poor quality of life) to 100 (maximum quality of life).
Time Frame: 6 months
Population: All participants who completed at 6 months were included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction (MBSR)
Number analyzed (Participants) | 65
units on a scale | 224.3 (96.3)

ADVERSE EVENTS:
Arm/Group | MBSR
Serious Adverse Events (participants affected / at risk) | 0/93
Other Adverse Events (participants affected / at risk) | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No